CLINICAL TRIAL: NCT04828538
Title: Prevent and Treat Double-Blind Factorial Randomized Trials of Daily Oral Vitamin D, Omega 3, and Combination Vitamins B, C and Zinc Supplementation for the Treatment and Prevention of COVID-19
Brief Title: Vitamin D, Omega-3, and Combination Vitamins B, C and Zinc Supplementation for the Treatment and Prevention of COVID-19
Acronym: NUTROVID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment failure
Sponsor: Hospital de la Soledad (Other Government)
Responsible Party: Principal Investigator, A Yáñez Admin, On-site Principal Investigator, Hospital de la Soledad
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 102020
Record Dates: First submitted 2021-03-12; First posted 2021-04-02 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: Covid19; Nutritional supplements; Vitamin B; Vitamin C; Elemental Zinc; Cytokine storm; Vitamin D; Vitamin B Complex; Omega 3
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Vitamin D; Ascorbic Acid; Vitamin B Complex; Zinc Acetate

STUDY DESIGN:
Intervention Model Description: Double-blind randomized, placebo-controlled double blinded 2x2x2 factorial trials (includes 2 trials: treatment cohort and prevention cohort) of the following oral supplementation treatments for up to 60 days per person:
  Factorial 1 (F1): 4000 IU Vitamin D vs placebo Factorial 2 (F2): 1000mg Omega DHA/EPA vs. placebo Factorial 3 (F3): Combination 1000 mg Vitamin C, Vitamin B complex** and Zinc Acetate, 100 mg/day vs. placebo
  **(Vitamin B complex components: B12=1 mg; B6=50 mg; B9=2.5 mg; B1
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 1 - Vitamin D, Omega 3, Vitamins B, C, Zinc (Active Comparator): Vitamin D of F1 Omega 3 of F2 Vitamins B, C, Zinc of F3
  [60 days]
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Omega DHA / EPA; Dietary Supplement: Vitamin C, Vitamin B complex and Zinc Acetate
- 2 - Vitamin D, Omega 3 (Active Comparator): Vitamin D of F1 Omega 3 of F2 Placebo of F3
  [60 days]
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Omega DHA / EPA
- 3 - Vitamin D, Vitamins B, C, Zinc (Active Comparator): Vitamin D of F1 Placebo of F2 Vitamins B, C, Zinc of F3
  [60 days]
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Vitamin C, Vitamin B complex and Zinc Acetate
- 4 - Vitamin D (Active Comparator): Vitamin D of F1 Placebo of F2 Placebo of F3
  [60 days]
  Interventions: Dietary Supplement: Vitamin D
- 5 - Omega 3, Vitamins B, C, Zinc, (Active Comparator): Placebo of F1 Omega 3 of F2 Vitamins B, C, Zinc of F3
  [60 days]
  Interventions: Dietary Supplement: Omega DHA / EPA; Dietary Supplement: Vitamin C, Vitamin B complex and Zinc Acetate
- 6 - Omega 3 (Active Comparator): Placebo of F1 Omega 3 of F2 Placebo of F3
  [60 days]
  Interventions: Dietary Supplement: Omega DHA / EPA
- 7 - Vitamins B, C, Zinc (Active Comparator): Placebo of F1 Placebo of F2 Vitamins B, C, Zinc of F3
  [60 days]
  Interventions: Dietary Supplement: Vitamin C, Vitamin B complex and Zinc Acetate
- 8 - No Interventions (Placebo Comparator): Placebo of F1 Placebo of F2 Placebo of F3
  [60 days]
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Daily 4000 IU Vitamin D for 60 days
  Arms: 1 - Vitamin D, Omega 3, Vitamins B, C, Zinc; 2 - Vitamin D, Omega 3; 3 - Vitamin D, Vitamins B, C, Zinc; 4 - Vitamin D
Dietary Supplement: Omega DHA / EPA — Daily 1000mg Omega DHA/EPA for 60 days
  Arms: 1 - Vitamin D, Omega 3, Vitamins B, C, Zinc; 2 - Vitamin D, Omega 3; 5 - Omega 3, Vitamins B, C, Zinc,; 6 - Omega 3
Dietary Supplement: Vitamin C, Vitamin B complex and Zinc Acetate — Combination 1000 mg Vitamin C, Vitamin B complex** and Zinc Acetate, 100 mg/day for 60 days
  **(Vitamin B complex components: B12=1 mg; B6=50 mg; B9=2.5 mg; B1=100 mg; B2=100 mg; B3=14 mg; B7=50 mg)
  Arms: 1 - Vitamin D, Omega 3, Vitamins B, C, Zinc; 3 - Vitamin D, Vitamins B, C, Zinc; 5 - Omega 3, Vitamins B, C, Zinc,; 7 - Vitamins B, C, Zinc
Other: Placebo — Placebo
  Arms: 8 - No Interventions

SUMMARY:
The NUTROVID Factorial Trials

The purpose of the NUTROVID-Prevent and NUTROVID-Treat Factorial Trials is to determine whether Vitamin B Complex, Vitamin C, and Zinc; Vitamin D; and Omega3, taken at dosages approximating recommended dosages, can reduce the risk of COVID-19 infection, hospitalization, mortality.

DETAILED DESCRIPTION:
Inadequate vitamin intake is common in Mexico. Vitamin deficiency is hypothesized as a risk factor for COVID-19 infection and severe outcomes. Specifically, Vitamin D has been hypothesized as a regulator of the inflammatory cytokine response; Vitamin C may help reduce the risk of a cytokine storm and support the immune system; Vitamin B reduces pro-inflammatory cytokine levels, helps improve respiratory function, reduces hypercoagulability, and promotes endothelial structural integrity; Resolvins, derived from Omega3s, are a type of specialized pro-resolving lipid autacoid mediators hypothesized to prevent cytokine storms. Elemental Zinc is hypothesized to inhibit the replication of viruses.

The NUTROVID-Prevent and NUTROVID-Treat Factorial Trials are testing the efficacy of these supplements (Vitamins B, C, D, Zinc, and Omega 3) when used over a 60 day period among those who test positive (Treat) and negative (Prevent) for SARS-COV-2 via a PCR test.

The NUTROVID Trials utilize an innovative and cost-efficient approach, leveraging the existing infrastructure of the hospital system in San Luis Potosí province of Mexico. For NUTROVID-Treat, we aim to enroll ~1,800 adults who have recently tested positive for SARS-Cov-2 and who have given informed consent. These ~1,800 adult females and males age 18 or older will be enrolled and randomized into the NUTROVID Treat Factorial Trial's 2x2x2 arms, in which 50% of the population will have a chance to receive any combination of the 3 supplement formulations; the other 50% will receive the respective placebos.

Those who test negative will be randomized into the NUTROVID-Prevent Factorial Trial's 2x2x2 arms, in which 50% of the population will have a chance to receive any combination of the 3 supplement formulations; the other 50% will receive the respective placebos. For NUTROVID-Prevent, we also aim to recruit ~1,800 adults, females and males.

Hospital staff will review medical records for vital events and conduct patient and family follow-up until ~November 2021.

ELIGIBILITY:
Positive SARS-CoV-2 Test group (Target enrollment: N=1,800) NUTROVID Treat Trial: Adult men/women recently diagnosed with COVID-19 (positive PCR test for SARS-CoV-2 coronavirus) within <=5 days of symptom onset; and satisfying one of these risk factors: >=50 years old; or Diabetic & >=40 years old; or Obese & >=40 years old.

Negative SARS-CoV-2 Test group (Target enrollment: N=1,800) NUTROVID Prevent Trial: Adult men/women recently tested negative for COVID-19 (negative PCR test for SARS-CoV-2 coronavirus); and satisfying one of these risk factors: >=50 years old; or Diabetic & >=40 years old; or Obese & >=40 years old.

Signed Informed Consent Form

Exclusion Criteria:

* Patients requiring immediate intubation or deemed likely to die within 48 hours.
* Patients deemed likely for transfer to an ICU within 48 hours.
* Patients currently taking oral corticosteroids for any reason at the time of presentation for care.
* Patients included in any other interventional trial.
* Uncontrolled bacterial superinfection.
* Severe chronic kidney disease (stage 4) or requiring dialysis (i.e. eGFR < 30).
* Pregnant women or women who are breastfeeding.
* Immunocompromised patients.
* Any patient with recent treatment (past 30 days) of immunosuppressive agents including (but not restricted to) DMARDs, corticosteroids, antibody therapy, intravenous immunoglobulins etc.
* Patients with acute myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Covid infection rate (PREVENT Trial only) | 30 and 60 days
  1.a. Incidence of positive PCR at ~1 month and ~2 months; 1.b. Incidence of symptomatic positive PCR and asymptomatic positive PCR at 1 month and 2 months.
Incidence of severe outcome (TREAT Trial only) | 1.a. 1-30 days; 1.b. 30-60; 1.c. 30 days to ~November 2021; 1.d. 60 days to ~ November 2021
  1.a. Incidence of severe outcome (mortality or ICU admission or intubation) up to 30 days.
  1.b. Incidence of severe outcome (mortality or ICU admission or intubation) from 30-60 days.
  1.c. Incidence of severe outcome (mortality or ICU admission or intubation), from 30 days to ~ November 2021.
  1.d. Incidence of severe outcome (mortality or ICU admission or intubation), from 60 days to
  ~ November 2021.

SECONDARY OUTCOMES:
Incidence of hospitalization and death (PREVENT Trial only) | 1-10 months
  2.a. Incidence of hospitalization, follow-up to ~ November 2021. 2.b. Incidence of severe outcome (mortality or ICU admission or intubation), follow-up to ~November 2021.
  2.c. Incidence of death, follow-up to ~November 2021.
Length of hospitalization and death after discharge (TREAT Trial only) | 2.a. 1-30 days; 2.b. 1 day(s) to ~November 2021, 2.c. 30 days to ~November 2021
  2.a. Length of hospitalization for admissions less than 30 days from baseline versus for admissions after 30 days from baseline. 2.b. [If available] Incidence of hospital readmission after discharge, follow-up to ~November 2021.
  2.c. Incidence of death after discharge, follow-up to ~November 2021.

OTHER OUTCOMES:
Changes in HbA1c (PREVENT Trial only) | 1-30; 1-60 days
  Change in HbA1c at 1 month and 2 months
Change in diabetes status (PREVENT Trial only) | 1-30; 1-60 days
  Change in diabetes status at 1 month and 2 months
Change in weight (PREVENT Trial only) | 1-30; 1-60 days
  Change in weight at 1 month and 2 months
Incidence of COVID -19 symptoms at 1 month and 2 months (PREVENT Trial only) | 1-30; 1-60 days
  [If available] Incidence of COVID -19 symptoms at 1 month and 2 months
Incidence of hospital readmission (PREVENT Trial only) | 1-30; 1-60 days; 1 day to ~November 2021
  [If available] Incidence of COVID -19 symptoms at 1 month and 2 months with follow-up to ~November 2021
Incidence of ICU admission (PREVENT Trial only) | 1-30; 1-60 days; 1 day to ~November 2021
  [If available] Incidence of ICU admission (PREVENT Trial only)
Incidence of intubation (PREVENT Trial only) | 1-30; 1-60 days; 1 day to ~November 2021
  [If available] Incidence of intubation (PREVENT Trial only)
Incidence of Vaccination (PREVENT Trial only) | 1-30; 1-60 days; 1 day to ~November 2021
  [If available] Incidence of vaccination
Change in HbA1c at 1 month and 2 months (TREAT Trial only) | 1-30 days and 1-60 days
  [If available] Change in HbA1c at 1 month and 2 months.
Change in diabetes status at 1 month and 2 months (TREAT Trial only) | 1-30 days and 1-60 days
  [If available] Change in diabetes status at 1 month and 2 months.
Change in weight at 1 month and 2 months (TREAT Trial only) | 1-30 days and 1-60 days
  [If available] Change in weight at 1 month and 2 months
Incidence of COVID -19 symptoms at 1 month and 2 months (TREAT Trial only) | 1-30 days and 1-60 days
  [If available] Incidence of COVID -19 symptoms at 1 month and 2 months.
Incidence of depression (TREAT Trial only) | ~1-60 days
  [If available] Incidence of depression
Incidence of vaccination (TREAT Trial only) | 1-30; 1-60 days; 1 day to ~November 2021
  [If available] Incidence of vaccination
Incidence of vaccine hesitancy (TREAT Trial only) | ~1-60 days
  [If available] Incidence of vaccine hesitancy
ICU readmission (TREAT Trial only) | 1-30; 1-60 days; 1 day to ~November 2021
  [If available] ICU readmission
Incidence of Intubation (upon readmission) (TREAT Trial only) | 1-30; 1-60 days; 1 day to ~November 2021
  [If available] Incidence of Intubation

CONTACTS AND LOCATIONS:
Overall Officials: José Yañez, Principal Investigator — General Hospital Soledad
Locations (1):
- Hospital de Soledad, San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Laird E, Rhodes J, Kenny RA. Vitamin D and Inflammation: Potential Implications for Severity of Covid-19. Ir Med J. 2020 May 7;113(5):81. PMID 32603576
- [Background] Boretti A, Banik BK. Intravenous vitamin C for reduction of cytokines storm in acute respiratory distress syndrome. PharmaNutrition. 2020 Jun;12:100190. doi: 10.1016/j.phanu.2020.100190. Epub 2020 Apr 21. PMID 32322486
- [Background] Panigrahy D, Gilligan MM, Huang S, Gartung A, Cortes-Puch I, Sime PJ, Phipps RP, Serhan CN, Hammock BD. Inflammation resolution: a dual-pronged approach to averting cytokine storms in COVID-19? Cancer Metastasis Rev. 2020 Jun;39(2):337-340. doi: 10.1007/s10555-020-09889-4. PMID 32385712
- [Background] Shakoor H, Feehan J, Mikkelsen K, Al Dhaheri AS, Ali HI, Platat C, Ismail LC, Stojanovska L, Apostolopoulos V. Be well: A potential role for vitamin B in COVID-19. Maturitas. 2021 Feb;144:108-111. doi: 10.1016/j.maturitas.2020.08.007. Epub 2020 Aug 15. No abstract available. PMID 32829981
- [Background] Entrenas Castillo M, Entrenas Costa LM, Vaquero Barrios JM, Alcala Diaz JF, Lopez Miranda J, Bouillon R, Quesada Gomez JM. "Effect of calcifediol treatment and best available therapy versus best available therapy on intensive care unit admission and mortality among patients hospitalized for COVID-19: A pilot randomized clinical study". J Steroid Biochem Mol Biol. 2020 Oct;203:105751. doi: 10.1016/j.jsbmb.2020.105751. Epub 2020 Aug 29. PMID 32871238
- [Background] Singh M, Das RR. Zinc for the common cold. Cochrane Database Syst Rev. 2013 Jun 18;(6):CD001364. doi: 10.1002/14651858.CD001364.pub4. PMID 23775705